CLINICAL TRIAL: NCT05541263
Title: 'MindRest: Mindful Network Dynamics Regulation Under Stress
Brief Title: Mindful Network Dynamics Regulation Under Stress
Acronym: MindRest
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was concluded early after including 75 participants, which fell short of our initial target of 120. This was mainly due to the impact of COVID-19 lockdowns and a higher than anticipated attrition rate.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL74345.091.20
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stress
Keywords: Mindfulness; Stress; Neuroimaging
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: We will perform a randomized, wait-list controlled trial with a Mindfulness-Based Stress Reduction (MBSR) intervention, based on the programme developed by Kabat-Zinn (1982).
Masking Description: Baseline Measurements will occur before group assignments and therefore both participants and researchers are blinded to these measurements. Post-treatment measurements are de-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBSR group (Experimental): The MBSR group participants will receive an Mindfulness Based Stress Reduction training programme over 2 months.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Wait-list group (No Intervention): The wait-list control group participants will wait while the experimental group is participating in the Mindfulness Based Stress Reduction training. This group will follow the training at the end of the study (7 months after baseline), after all relevant measurements are concluded.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — The intervention used is an MBSR training which is based on the Mindfulness-Based Stress Reduction programme as developed by Kabat-Zinn (1982). The training consists of 8 weekly sessions lasting 2,5 hours. A silent day of approximately 6 hours is also included, as well as daily home practice assignments of about 45 minutes. During the training participants will learn to focus their attention in the present moment in an accepting and non-judgemental way, rather than ruminating about past and future experiences. The training includes formal exercises during which participants will practice the body scan, sitting meditation, walking meditation and mindful movement. Informal exercises are also included, such as performing a daily activity with full attention to the present experience. The training is led by qualified teachers meeting the advanced criteria of the Association of Mindfulness Based Teachers in the Netherlands and Flanders (www.vmbn.nl)
  Other Names: MBSR
  Arms: MBSR group

SUMMARY:
This study aims to assess the effectiveness of Mindfulness Based Stress reduction to reduce perceived stress in a highly stressed student population, while concurrently investigating neural mechanisms of the intervention. The investigators will perform a randomized, wait-list controlled trial assessing clinical and neurocognitive outcomes as well as measures of daily life stress reactivity.

DETAILED DESCRIPTION:
Rationale: Prolonged stress exposure can put people at risk of developing stress-related symptomatology, such as burnout, sleeping disorders, depression and anxiety. Students reporting high levels of perceived stress are an at-risk population that could potentially benefit from a stress-reduction intervention. One approach to reduce stress is Mindfulness Based Stress Reduction (MBSR). Although proven effective, additional evidence is required on the effectiveness of MBSR in reducing stress-related symptoms in student sample pre-selected on high stress. Furthermore, the working mechanisms of MBSR are only marginally understood. This is problematic, because gaining better mechanistic insight on how MBSR works might lead (1) to basic scientific insights into stress and stress resilience and (2) clinically, to improve the provided interventions . In the light of preliminary psychological study results on MBSR the investigators hypothesize that MBSR will not only foster stress-reduction via cognitive control but also via experiential exposure. In accordance with this hypothesis and based on neurocognitive findings in basic stress research and previous mechanistic studies on MBSR, the investigators will assess whether MBSR indeed leads to improved stress-regulation by enhancing both cognitive and affective processing, which will be reflected in neural network configuration.

Objective: The main objective of this study is to assess the effectiveness of MBSR to reduce perceived stress in a highly stressed student population. Our main objective regarding working mechanisms of MBSR is to assess possible MBSR induced changes in large-scale neural network configuration and self-regulation of these networks. Additionally, this study aims to explore possible mediators and moderators of the treatment effect, both in terms of psychological traits, and neural patterns.

Study design: The investigators will perform a two-arm randomized, wait-list controlled trial with a randomisation ratio of 1:1. Participants will be randomised into a treatment and wait-list group after baseline Clinical Assessments (CA), Neurocognitive Assessments (NA), and Ecological Momentary Assessments (EMA). In the following two months the experimental group will participate in an MBSR training and the control group will wait for two months. Another CA and NA and EMA will take place 3 months after baseline. 6 months after baseline there will be a follow-up CA. Participants in the wait-list group will then receive an MBSR training, after which they will perform another CA.

Study population: The investigators will recruit 60 students per group ( total: 120) from Radboud University, Radboudumc, and HAN University of Applied Sciences in Arnhem and Nijmegen with high perceived stress. Participants above 18 years, able to give consent, who score ≥ 16 on the Perceived Stress Scale will be prompted to join our study. Participants will be excluded if they are receiving current specialised psychological or psychiatric treatment or medication, if they have insufficient comprehension of the Dutch language, if they have physical, cognitive, or intellectual impairments interfering with participation, such as deafness, blindness, or sensori-motor handicaps, if they were formerly or currently involved in MBCT or MBSR training, if they have a current drug or alcohol addiction, and if they have contraindications for MRI scanning (e.g., pacemaker, implanted metal parts, deep brain stimulation, claustrophobia, epilepsy, brain surgery, pregnancy).

Intervention: Participants in the treatment group will follow an MBSR training which consists of 8 weekly sessions lasting 2,5 hours; a silent day of approximately 6 hours; and daily home practice assignments of about 45 minutes. The control group will follow the training at the end of the study (7 months after baseline), therefore acting as a wait-list control group during the measurements.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent.
* Perceived Stress Scale score ≥ 16.

Exclusion Criteria:

* Current specialised psychological or psychiatric treatment or medication.
* Insufficient comprehension of the Dutch language.
* Physical, cognitive, or intellectual impairments interfering with participation, such as deafness, blindness, or sensori-motor handicaps.
* Formerly/currently involved in MBCT or MBSR training.
* Current drug or alcohol addiction.
* Contraindications for MRI scanning (e.g., pacemaker, implanted metal parts, deep brain stimulation, claustrophobia, epilepsy, brain surgery, pregnancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Difference in perceived stress between experimental and control group | Change between baseline and 3 months
  This is measured by the total score of the Perceived Stress Scale (PSS) 10-item questionnaire (range 0-40), which evaluates the degree to which an individual perceives their life as unpredictable, uncontrollable and overloading.

SECONDARY OUTCOMES:
Depressive symptoms | At baseline, 3 months, 6 months
  Assessed with the IDS-SR: Inventory of Depressive Symptomatology Self-Report, which is a self-reported 30-item measure of depressive symptom severity (range 0-93).
Anxiety | At baseline, 3 months, 6 months
  Assessed with the STAI: State and Trait Anxiety Inventory, which is a self-reported 20-item measure of trait (range 20-80) and a self-reported 20-item measure (range 20-80) state anxiety.
Alcohol use | At baseline, 3 months, 6 months
  Assessed with the AUDIT: Alcohol Use Disorders Identification Test, which is a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, drinking behaviours, and alcohol-related problems (range 0-40).
Childhood trauma | At baseline
  Assessed with the MACE-X: Maltreatment and Abuse Chronology of Exposure Scale, which is a self-reported questionnaire which used to assess the extent as well as the severity of traumatic experiences of participants in their childhood.
Personality traits | At baseline, 3 months, 6 months
  Assessed with the NEO-FFI: NEO Five Factor Inventory, which is a 60-item self-reported questionnaire and covers a set of five broad personality trait dimensions or domains: Extraversion, Agreeableness, Conscientiousness, Neuroticism, and Openness to Experience.
Repetitive negative thinking | At baseline, 3 months, 6 months
  Assessed with the PTQ: Perseverative Thinking Questionnaire, which is a 15-item self-reported questionnaire and is used to assess repetitive negative thinking in a content-free manner (range 0-60).
Cognitive reactivity | At baseline, 3 months, 6 months
  Assessed with the LEIDS-R: Leiden Index of Depression Sensitivity - Revised, which is a 34-item self-reported questionnaire measuring cognitive reactivity to sadness (range 0-136).
Allowing of emotions | At baseline, 3 months, 6 months
  Assessed with the AAQ: Acceptance and Action Questionnaire, which is a 10-item self-reported questionnaire measuring psychological flexibility and experiential acceptance (range 10-70).
Mindfulness skills | Time Frame: At baseline, 3 months, 6 months
  Assessed with the FFMQ-SF: short version of the Five-Facet Mindfulness Questionnaire, which is a 24-item self-reported questionnaire measuring five aspects of mindfulness, namely observation, description, aware actions, non-judgemental inner experience, and non-reactivity.
Self-compassion | At baseline, 3 months, 6 months
  Assessed with the SCS-S: short version of the Self-Compassion Scale, which is a 12-item self-reported questionnaire measuring consisting of six components, including self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification.
Stress Resilience | At baseline, 3 months, 6 months
  Assessed with the CD-RISC: Connor-Davidson Resilience Scale, which is a 25-item self-reported measure of stress resilience (range 0-100)
Positive mental health | At baseline, 3 months, 6 months
  Assessed with the MHC-SF: short form of the Mental Health Continuum, which is a 14-item self-report questionnaire that assesses emotional, psychological and social well-being (range 0-70).
Blood Oxygen Level Dependent (BOLD) signal | At baseline, 3 months
  Assessed using Functional Magnetic Resonance Imaging (fMRI) during four tasks (Resting State, Fear conditioning paradigm, Emotional Stroop task, and Self-regulation using neurofeedback). This will be used to determine activity, connectivity and cohesion patterns of largescale brain networks during these stress regulation tasks.
Automatic exogenous stress regulation | At baseline, 3 months
  Assessed using a differential fear conditioning and extinction paradigm. This task will be used to measure the retention of safety learning in an experimental model of exposure therapy. This measure is operationalized as the reduction of spontaneous recovery of autonomic nervous system reactivity (skin conductance, heart rate, and pupil dilation responses) to fear-conditioned stimuli one day after extinction of fearful memories (i.e., safety learning).
Controlled exogenous stress regulation | At baseline, 3 months
  Assessed during a Stroop-like emotional conflict resolution task. We will measure cognitive control processes in the context of conflicting emotional information by measuring reaction times and accuracy scores during the task.
Automatic endogenous stress regulation | At baseline, 3 months
  Assessed using during a resting state Functional Magnetic Resonance Imaging (fMRI) scan following a laboratory stress-induction procedure. Stress responses will be assessed through repeated measurement of salivary cortisol levels, pupillary responses and heart rate.
Controlled endogenous stress regulation | At baseline, 3 months
  Assessed using a Real-time Functional Magnetic Resonance Imaging (fMRI) Neurofeedback task based on largescale brain network balance. This task will test individuals' ability to dynamically self-regulate their configuration of largescale brain networks.

OTHER OUTCOMES:
Daily life stress reactivity | At baseline, 3 months
  Assessed using 6 surveys per day with mood- and stress-related questions (i.e. ecological momentary assessments) for 6 continuous days, coupled with physiological measures (heart rate, skin conductance, skin temperature, and movement), to assess stress reactivity in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Erno Hermans, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon request using the Donders Institute research data repository (http://data.donders.ru.nl) in accordance to institutional and EU guidelines.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will be stored and archived through the data management infrastructure of the Donders Institute, and will be kept for at least 15 years.
Access Criteria: Access to data is managed by the researchers responsible for the data and they can decide to give access rights to other individuals when necessary or requested.

REFERENCES:
- [Background] Alsubaie M, Abbott R, Dunn B, Dickens C, Keil TF, Henley W, Kuyken W. Mechanisms of action in mindfulness-based cognitive therapy (MBCT) and mindfulness-based stress reduction (MBSR) in people with physical and/or psychological conditions: A systematic review. Clin Psychol Rev. 2017 Jul;55:74-91. doi: 10.1016/j.cpr.2017.04.008. Epub 2017 Apr 23. PMID 28501707
- [Background] Hermans EJ, Henckens MJ, Joels M, Fernandez G. Dynamic adaptation of large-scale brain networks in response to acute stressors. Trends Neurosci. 2014 Jun;37(6):304-14. doi: 10.1016/j.tins.2014.03.006. Epub 2014 Apr 21. PMID 24766931
- [Background] Lyndon MP, Strom JM, Alyami HM, Yu TC, Wilson NC, Singh PP, Lemanu DP, Yielder J, Hill AG. The relationship between academic assessment and psychological distress among medical students: a systematic review. Perspect Med Educ. 2014 Dec;3(6):405-418. doi: 10.1007/s40037-014-0148-6. PMID 25428333
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Derived] Kogias N, Geurts DEM, Krause F, Speckens AEM, Hermans EJ. Study protocol for a randomised controlled trial investigating the effects of Mindfulness Based Stress Reduction on stress regulation and associated neurocognitive mechanisms in stressed university students: the MindRest study. BMC Psychol. 2023 Jul 1;11(1):194. doi: 10.1186/s40359-023-01220-4. PMID 37393359